CLINICAL TRIAL: NCT01861002
Title: A Phase I Study of 5-Azacytidine in Combination With Chemotherapy for Children With Relapsed or Refractory ALL or AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2011-002
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood; Myelogenous Leukemia, Acute, Childhood
Keywords: Relapse; Lymphoblastic; Leukemia; Azacytidine; Refractory; Myelogenous; Acute; Childhood; Pediatric; ALL; AML; Methylation; Epigenetic therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid; Recurrence; Leukemia | interventions — Azacitidine; fludarabine; fludarabine phosphate; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AML Arm (Experimental): Participants with Acute Myeloid Leukemia (AML)
  Intervention:
  * Azacytidine (Dose Level 1 @ 75 mg/m2/day)
  * Fludarabine 30 mg/m2/dose
  * Cytarabine 2000 mg/m2/dose
  * Intrathecal (IT) Cytarabine
  Interventions: Drug: Azacytidine; Drug: Fludarabine; Drug: Cytarabine; Drug: Intrathecal (IT) Cytarabine
- ALL Arm (Experimental): Patients with Acute Lymphocytic Leukemia
  Intervention:
  * Azacytidine (Dose Level 1 @ 75 mg/m2/day)
  * Fludarabine 30 mg/m2/dose
  * Cytarabine 2000 mg/m2/dose
  * Intrathecal Methotrexate (IT MTX)
  Interventions: Drug: Azacytidine; Drug: Fludarabine; Drug: Cytarabine; Drug: Intrathecal Methotrexate (IT MTX)

INTERVENTIONS:
Drug: Azacytidine — Dose assigned at study entry (75 mg/m2/day). Given subcutaneously, once daily on days 1 to 5, for a total of 5 doses.
  Other Names: 5 Azacytidine; Vidaza
Drug: Fludarabine — 30 mg/m2/dose, intravenous infusion over 30 minutes, once daily, on days 6 to 10, total 5 doses
  Other Names: fludarabine phosphate; Fludara; 2-fluoro-ara-AMP; Oforta
Drug: Cytarabine — 2000 mg/m2/dose intravenous infusion over 3 hours, starting 4 hours after the beginning of fludarabine, once daily, on days 6 to 10, total 5 doses.
  Other Names: Cytosar-U; Ara-C; Arabinosylcytosine; cytosine arabinoside
Drug: Intrathecal (IT) Cytarabine — Intrathecally to AML patients on day 1 of course 1 and 2.
  * Omit on day 1 of course 1 if patient received IT therapy within 7 days prior to study enrollment
  * IT therapy may be given during the end of course 1 disease evaluation and repeated every 7 days
  * For patients with CNS disease, IT cytarabine can be given weekly until the CSF is clear. Two additional doses of IT cytarabine should be given weekly after the initial CSF clearing. It is permitted to change to intrathecal triple therapy (ITT) if persistent blasts are present in the CSF based on the treating physician's clinical judgment. Cytarabine dose defined by age:
  * 30 mg for patients age 1-1.99
  * 50 mg for patients age 2-2.99
  * 70 mg for patients >3 years of age
  ITT Dosing:
  Age (yrs) - Dose Methotrexate (MTX), Hydrocortisone (HC), Cytarabine (ARAC):
  1. - 1.99 MTX: 8 mg, HC: 15 mg, ARAC: 30 mg
  2. - 2.99 MTX: 10 mg, HC: 25 mg, ARAC: 50 mg
     * 3 - MTX: 12 mg, HC: 35 mg, ARAC: 70 mg
  Other Names: (See Cytarabine)
  Arms: AML Arm
Drug: Intrathecal Methotrexate (IT MTX) — * Intrathecally to patients with ALL on day 1 of course 1 and 2.
  * Omit IT MTX on Day 1 of course 1 if patient received IT therapy within 7 days prior to study enrollment
  * IT therapy may be given during the end of course 1 disease evaluation and repeated every 7 days
  * For patients with CNS 2 or 3 disease, IT MTX can be given weekly until the CSF is clear. Two additional doses of IT MTX should be given weekly after the initial clearing of the CSF. It is permitted to change to ITT if persistent blasts are present in the CSF. Methotrexate dose defined by age
  * 8 mg for patients age 1-1.99
  * 10 mg for patients age 2-2.99
  * 12 mg for patients 3-8.99 years of age
  * 15 mg for patients >9 years of age
  Triple IT Therapy Dosing:
  Age (yrs): Dose Methotrexate (MTX), Hydrocortisone (HC), Cytarabine (ARAC):
  1. - 1.99 MTX: 8 mg, HC: 8 mg, ARAC: 16 mg
  2. - 2.99 MTX: 10 mg, HC: 10 mg, ARAC: 20 mg
  3. - 8.99 MTX: 12 mg, HC: 12 mg, ARAC: 24 mg
     * 9 MTX: 15 mg, HC: 15 mg, ARAC: 30 mg
  Other Names: Otrexup; Rasuvo; Rheumatrex; Trexall; Amethopterin; Methotrexate Sodium
  Arms: ALL Arm

SUMMARY:
This is a Phase I study with a conditional cohort expansion phase to evaluate the feasibility of, and to obtain preliminary efficacy data about, pretreatment with Azacytidine (AZA) for 5 days followed by fludarabine/cytarabine chemotherapy regimen in pediatric acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL) patients who are refractory to primary treatment or who relapsed.

DETAILED DESCRIPTION:
Growing evidence indicates that aberrant DNA hypermethylation is associated with leukemia development, drug resistance, and relapse. It has been shown that pretreating leukemia cells with AZA or decitabine could partially reverse the aberrant DNA methylation, restore the expression of tumor suppressor gene important for apoptosis, and sensitize cells to subsequent killing by cytotoxic agent. Since cytarabine and decitabine share the same mechanisms of resistance, we use AZA to test the novel epigenetic "priming" approach. This is a phase I clinical study with expansion phase, using hypomethylating agent, 5-azacytidine (AZA), in sequential with chemotherapy to evaluate whether epigenetic "priming" can reverse aberrant DNA methylation, overcome drug resistance, and increase response in relapsed/refractory AML.

The chemotherapy regimen to be used in this study is fludarabine and cytarabine. This regimen has substantial activity in leukemia and has been widely used in treating pediatric patients with relapsed/refractory AML and ALL in the past several decades. In BFM relapsed AML 2001/01 study, FLAG (fludarabine, cytarabine and G-CSF) chemotherapy regimen showed significant activity in AML with 4 year OS around 36%. Since the use of G-CSF in conjunction with fludarabine/cytarabine didn't improve the overall survival of patient in a randomized trial, only fludarabine and cytarabine will be used in this study to decrease the incidence of leukocytosis related complications. This regimen is very similar to the chemotherapy regimen proposed for the next relapsed AML trial within the Children's Oncology Group (COG). If this trial proves to be safe and active, it will provide the foundation and smooth transition to larger statistically powered nationwide phase II clinical trials by COG.

ELIGIBILITY:
Inclusion Criteria:

Patients must be ≥ 1 and ≤ 21 years of age.

Diagnosis

1. Patients with AML must have ≥5% blasts (by morphology) in the bone marrow.
2. Patients with ALL must have an M2 or M3 marrow (≥5% blasts by morphology).
3. Patients may have disease in the central nervous system (CNS) or other sites of extramedullary disease. No cranial irradiation is allowed during the protocol therapy.
4. Patients with secondary AML are eligible.
5. Patients with Down syndrome and DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome) are excluded.

Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients ≤ 16 years of age.

Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

Myelosuppressive chemotherapy - the eligibility criteria is different between phase I and expansion phase

1. Phase I

   * Any patient with AML in 1st or greater relapse, OR
   * Any patient with ALL in 2nd or greater relapse, OR
   * Patients with AML or ALL failed to go into remission after first or greater relapse, OR
   * Patients with AML or ALL failed to go into remission from original diagnosis after two or more courses of induction attempts.
2. Expansion phase - will be restricted to AML patients only
3. Cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of azacytidine. It is recommended to use hydroxyurea in patients with significant leukocytosis (WBC > 50,000/L) to control blast count before initiation of systemic protocol therapy.
4. Patients who relapsed while they are receiving cytotoxic therapy (including AZA , decitabine, or vorinostat) At least 14 days must have elapsed since the completion of the cytotoxic therapy.

Hematopoietic stem cell transplant: Patients who have experienced their relapse after a stem cell transplant are eligible, provided they have no evidence of acute or chronic Graft-versus-Host Disease (GVHD) and are at least 90 days post-transplant at the time of enrollment.

Hematopoietic growth factors: It must have been at least 7 days since the completion of therapy with filgrastim or other growth factors at the time of enrollment. It must have been at least 14 days since the completion of therapy with pegfilgrastim (Neulasta®).

Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair

Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of monoclonal antibody. (i.e. Gemtuzumab = 36 days)

Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.

Radiation Therapy (XRT): Craniospinal XRT is prohibited during protocol therapy. No washout period is necessary for radiation given to non-CNS chloromas; ≥ 90 days must have elapsed if prior total body radiation or craniospinal radiation.

Renal and hepatic function

Patients must have adequate renal and hepatic functions as indicated by the following laboratory values:

* Patient must have a calculated creatinine clearance or radioisotope glomerular filtration rate (GFR) greater than or equal to 70ml/min/1.73m2 OR a normal serum creatinine based on age/gender.
* Direct bilirubin < 1.5 x upper limit of normal (ULN) for age or normal, AND alanine transaminase (ALT) < 5 x ULN for age.

Adequate Cardiac Function Defined as: Shortening fraction greater than or equal to 27% by echocardiogram, OR ejection fraction greater than or equal to 50% by radionuclide angiogram (MUGA).

Reproductive Function

* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 2 weeks prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.

Patients and/or their parents or legal guardians must be capable of understanding the investigational nature, potential risks and benefits of the study. All patients and/or their parents or legal guardians must sign a written informed consent.

Exclusion Criteria:

Patients will be excluded if they have a known allergy to any of the drugs used in the study.

Patients will be excluded if they have a systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient needs to be off pressors and have negative blood cultures for 48 hours.

Patients will be excluded if there is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.

Patients will be excluded if they have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results.

Patients with Down syndrome and DNA fragility syndromes (such as Fanconi anemia, Bloom syndrome) are excluded.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05-22 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2014-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weili Sun, MD, PhD, Study Chair — Children's Hospital Los Angeles
Locations (23):
- United States (19):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCSF School of Medicine, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Emory University, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber, Boston, Massachusetts
  - C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Childrens Hospital & Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Hospital New York-Presbyterian, New York, New York
  - Levine Children's Hospital at Carolinas Medical Center, Charlotte, North Carolina
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Texas at Southwestern, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Children's Hospital at Westmead, Westmead, New South Wales
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Sainte-Justine University Hospital Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun W, Triche T Jr, Malvar J, Gaynon P, Sposto R, Yang X, Bittencourt H, Place AE, Messinger Y, Fraser C, Dalla-Pozza L, Salhia B, Jones P, Wayne AS, Gore L, Cooper TM, Liang G. A phase 1 study of azacitidine combined with chemotherapy in childhood leukemia: a report from the TACL consortium. Blood. 2018 Mar 8;131(10):1145-1148. doi: 10.1182/blood-2017-09-803809. Epub 2018 Jan 16. No abstract available. PMID 29339403
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- 75 mg/m2/Day Azacytidine: * Azacytidine (Dose Level @ 75 mg/m2/day),all patients will start at Dose Level 1. If 2 DLTs are observed within the first 6 patients enrolled, dose will be reduced to Dose Level 0 @ 50 mg/m2/day
  * Fludarabine 30 mg/m2/dose
  * Cytarabine 2000 mg/m2/dose
  * Intrathecal (IT) Cytarabine
Period: Overall Study
Arm/Group | 75 mg/m2/Day Azacytidine
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Number that completed therapy and were analyzed
Groups:
- Dose Level 1 75 mg/m2/Day: This arm is comprised of the AML and ALL participants that completed Dose Level 1 75 mg/m2/day
Arm/Group | Dose Level 1 75 mg/m2/Day
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 9.7 [1.4 to 16.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Central Nervous System (CNS) Status [Count of Participants; unit: Participants] — CNS Negative (better outcome): absence of blasts on a cytospin preparation in cerebral spinal fluid (CSF) or clinical signs of CNS leukemia
  CNS Positive (worse outcome): presence of any number of blasts on a cytospin preparation in CSF or clinical signs of CNS leukemia
  Participants
    CNS Negative | 8
    CNS Positive | 6
Bone Marrow Status (at study entry) [Count of Participants; unit: Participants] — Measurement of bone marrow response
  M2 (better outcome): Marrow has between 5% and 25% leukemic blasts M3 (worse outcome): Marrow has more than 25% leukemic blasts
  Participants
    M2 (5-25% Leukemic Blasts) | 5
    M3 (>25% Leukemic Blasts) | 9
# Prior treatment regimens [Count of Participants; unit: Participants]
  1 prior treatment | 4
  2 prior treatments | 4
  3 or more prior treatments | 6
Prior Hematopoetic Stem Cell Transplantation (HSCT) [Count of Participants; unit: Participants]
  No Previous HSCT | 9
  Previous HSCT | 5
White blood cell (WBC) Count [Median (Full Range); unit: Thousand cells / mm^3] | 6.89 [0.61 to 49.9]
Peripheral blasts [Median (Full Range); unit: Percentage of cells] | 16 [0 to 86]
Bone marrow blasts [Median (Full Range); unit: Percentage of cells] | 68.5 [16 to 94]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose Limiting Toxicity (DLT)
Description: To evaluate the side effects of giving Azacytidine before and during chemotherapy using the standard drugs Fludarabine, Cytarabine, IT Cytarabine (AML patients) and IT methotrexate (ALL patients)
Time Frame: From Day 1 to Day 42 (Cycle 1)
Measure: Count of Participants; unit: Participants
Groups:
- Dose 75 mg/m2/Day Azacytidine Diagnosed With AML: Evaluable Participants who received azacytidine @ 75 mg/m2/day (Dose Level 1)
- Dose 75 mg/m2/Day Azacytidine Diagnosed With ALL: Evaluable ALL participants who received azacytidine @ 75 mg/m2/day (Dose Level 1)
Arm/Group | Dose 75 mg/m2/Day Azacytidine Diagnosed With AML | Dose 75 mg/m2/Day Azacytidine Diagnosed With ALL
Number analyzed (Participants) | 13 | 2
Participants
  # of patients with DLT | 0 | 0
  # of patients without DLT | 12 | 2
  # of patients not evaluable | 1 | 0

2. Secondary Outcome: Disease Response Rate After Treatment
Description: CR is defined as a bone marrow with < 5% blast by morphology, no evidence of extramedullary disease, and recovery of peripheral counts (ANC ≥ 1000/μl and platelet counts ≥ 100,000/μl). CR with incomplete count recovery (CRi) was defined as CR without recovery of ANC and/or platelets. Partial response (PR) was defined as complete disappearance of circulating blasts and a decrease of at least 50% of blasts in the bone marrow. Progressive disease (PD) was defined as an increase of at least 25% in the absolute number of bone marrow or circulating blasts, development of new sites of extramedullary disease, or other laboratory or clinical evidence of progression of disease. Stable disease (SD) referred to patient who did not satisfy the criteria for either CR, CRi, PR or PD.
Time Frame: Between Days 36-42 of Courses 1 and 2
Measure: Count of Participants; unit: Participants
Groups:
- Dose 75 mg/m2/Day for AML Patients: Participants with Acute Myeloid Leukemia (AML) who are evaluable for response.
  A patient will be considered evaluable for response if: (1) the patient is eligible; (2) the patient receives all or part of protocol therapy; and (3) the patient is under follow-up for a sufficient period to evaluate the disease at the end of the course 2 or meets the definition of progressive disease. A patient who dies as a result of toxicity after receiving all or part of protocol therapy will be considered a non-responder.
  Intervention:
  * Azacytidine (Dose Level 1 @ 75 mg/m^2/day)
  * Fludarabine 30 mg/m^2/dose
  * Cytarabine 2000 mg/m^2/dose
  * Intrathecal (IT) Cytarabine
- Dose 75 mg/m2/Dose Azacytidine for ALL Patients: Participants with Acute Lymphoblastic Leukemia (ALL) who are evaluable for response.
  A patient will be considered evaluable for response if: (1) the patient is eligible; (2) the patient receives all or part of protocol therapy; and (3) the patient is under follow-up for a sufficient period to evaluate the disease at the end of the course 2 or meets the definition of progressive disease. A patient who dies as a result of toxicity after receiving all or part of protocol therapy will be considered a non-responder.
  Intervention:
  * Azacytidine (Dose Level 1 @ 75 mg/m^2/day)
  * Fludarabine 30 mg/m^2/dose
  * Cytarabine 2000 mg/m^2/dose
  * Intrathecal (IT) Methotrexate
Arm/Group | Dose 75 mg/m2/Day for AML Patients | Dose 75 mg/m2/Dose Azacytidine for ALL Patients
Number analyzed (Participants) | 12 | 2
Participants
  Complete Remission (CR) | 6 | 0
  CR with Incomplete Count Recovery (CRi) | 1 | 0
  Partial Remission (PR) | 1 | 1
  Stable Disease (SD) | 1 | 1
  Progressive Disease (PD) | 3 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose of AZA until 30 days following the last dose of protocol therapy (approximately from Day 0 to Day 112)
Description: The definitions of AE and SAE do not differ from the clinicaltrials.gov definitions.
Groups:
- AML Cohort: 75 mg/m2/Day: Any patients in the AML arm who are evaluable for toxicity. Any patient who experiences a DLT after receiving at least one dose of AZA on study will be considered evaluable for toxicity of AZA. Patients who do not experience a DLT must receive at least 80% of the prescribed course of AZA in the first cycle (i.e., must receive at least 4 of the planned 5 doses of AZA between days 1 to 5) to be evaluable for toxicity of AZA. Patients not evaluable for toxicity of AZA will be replaced.
- ALL Cohort: 75 mg/m2/Day: Any patients in the ALL arm who are evaluable for toxicity. Any patient who experiences a DLT after receiving at least one dose of AZA on study will be considered evaluable for toxicity of AZA. Patients who do not experience a DLT must receive at least 80% of the prescribed course of AZA in the first cycle (i.e., must receive at least 4 of the planned 5 doses of AZA between days 1 to 5) to be evaluable for toxicity of AZA. Patients not evaluable for toxicity of AZA will be replaced.
Arm/Group | AML Cohort: 75 mg/m2/Day | ALL Cohort: 75 mg/m2/Day
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/2
Serious Adverse Events (participants affected / at risk) | 5/13 | 1/2
Other Adverse Events (participants affected / at risk) | 13/13 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AML Cohort: 75 mg/m2/Day (N=13) | ALL Cohort: 75 mg/m2/Day (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Fever (General disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 2 | 0 — 1 patient: Blood culture taken from central line positive for Klebsiella pneumoniae 1 patient: E. Coli Sepsis
Sepsis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AML Cohort: 75 mg/m2/Day (N=13) | ALL Cohort: 75 mg/m2/Day (N=2)
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 0
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 11 | 1
Alkaline phosphatase increased (Investigations) | 2 | 0
Allergic reaction (Immune system disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Anal pain (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 10 | 2
Anorexia (Metabolism and nutrition disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 11 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Blood bilirubin increased (Investigations) | 4 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 5 | 0
Chills (General disorders) | 1 | 0
Cholesterol high (Investigations) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Creatinine increased (Investigations) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 0
Dizziness (Nervous system disorders) | 3 | 0
Dry eye (Eye disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Edema face (General disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 — Bilateral eye irritation
Eye pain (Eye disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 2
Fever (General disorders) | 10 | 0
Fibrinogen decreased (Investigations) | 1 | 0
GGT increased (Investigations) | 3 | 0
Headache (Nervous system disorders) | 4 | 0
Hematuria (Renal and urinary disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 7 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 13 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatremia (Metabolism and nutrition disorders) | 6 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 0
Hypotension (Vascular disorders) | 1 | 1
Infections and infestations - Other, specify (Infections and infestations) | 4 | 1 — Various: Klebsiella pneumoniae; Epstein Barr; Enterococci; HSV, E. Coli; clostridium difficile; streptococcus sanguis; rhinovirus; Anchromobacter dentrificans
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Infusion site extravasation (Injury, poisoning and procedural complications) | 2 | 0
Injury, poisoning & proc complications - Other (Injury, poisoning and procedural complications) | 1 | 0 — Penis Laceration
INR increased (Investigations) | 2 | 0
Investigations - Other, specify (Investigations) | 2 | 0 — Hypochloremia; bicarbonate serum low; hemoptysis
Irritability (Psychiatric disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 | 0 — Chloride level decreased
Mucosal infection (Infections and infestations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 4 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 3 | 0 — Altered mental status; related to Benadryl; night terrors; pupillary dilation related to scopolamine, Altered mental status, cytarabine related
Neutrophil count decreased (Blood and lymphatic system disorders) | 11 | 1
Non-cardiac chest pain (General disorders) | 3 | 0
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Erythema & Swelling (Skin and subcutaneous tissue disorders) | 1 | 0
Gum Bleeding (Gastrointestinal disorders) | 1 | 0
Pain (General disorders) | 6 | 0 — Pain related to refractory Chloromas, Throat Pain. Epigastric Pain, Painful Urination, abdominal pain at time of physical exam, pain at site of injection, pain at the site of injection of azacytidine, pain left shoulder related to aza or picc line
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Photophobia (Eye disorders) | 1 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 12 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory, thoracic & mediastinal disorder-Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Serum amylase increased (Investigations) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 3 | 0
Skin & subcutaneous tissue disorder-Other (Skin and subcutaneous tissue disorders) | 6 | 0 — Skin rash or injection site redness after administration of 5 aza (N=5); Celullitis; Lower Extremity Rash; Dry Lips; Blister, Right Upper Extremity; burning sensation to scalp; anal fissure; skin rash following administration of vancomycine
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 2 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 0
Weight gain (Metabolism and nutrition disorders) | 1 | 0
Weight loss (Metabolism and nutrition disorders) | 2 | 0
White blood cell decreased (Investigations) | 11 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days